CLINICAL TRIAL: NCT00847509
Title: A Phase II/III, Open Label, Non-Randomized, Multi - Center Study Of Positron Emission Tomography (PET) Imaging With [F-18] FLT Compared to [F-18] FDG in Cancer Patients for Treatment Evaluation
Brief Title: A Multi - Center Study Of PET Imaging With [F-18] FLT & [F-18] FDG in Cancer Patients for Treatment Evaluation
Acronym: FLT101
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Siemens Molecular Imaging (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FLT101
Record Dates: First submitted 2009-02-17; First posted 2009-02-19 (Estimated); Results first posted 2013-09-27 (Estimated); Last update posted 2013-09-27 (Estimated); Status verified 2013-07

CONDITIONS: Lung Cancer; Head and Neck Cancer
Keywords: lung cancer; head and neck cancer; radiotherapy; chemoradiotherapy; radiation; chemoradiation; FLT; [F-18]FLT; FDG; [F-18]FDG
MeSH Terms: conditions — Lung Neoplasms; Head and Neck Neoplasms | interventions — alovudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FLT PET scan (Experimental): Open label, nonrandomized, uncontrolled, single group assignment, multi-center clinical trial to evaluate [F-18] FLT as a PET imaging tool in cancer patients clinically scheduled for treatment with radiation or radiation - chemotherapy. Standard [F-18] FDG PET will be the active comparator.
  Interventions: Drug: [F-18]FLT

INTERVENTIONS:
Drug: [F-18]FLT — The individual doses of [F-18]FLT contain a maximum of 10 mCi. The single IP dose is administered to the study subject approximately 30 to 60 minutes prior to the start of PET imaging.
  Other Names: [F-18] FLT; FLT

SUMMARY:
Approximately 60 patients will be enrolled with highly suspected lung cancer, or head and neck cancer. The patients must also be starting radiotherapy or a chemoradiotherapy regimen (except with 5-fluorouracil). The patients will undergo 3 visits. One screening, one pre therapy PET/CT imaging visit, and one (3-5 weeks after the start of therapy) post PET/CT imaging visit. This study will evaluate the FLT and FDG images for tumor proliferation rates for early assessment of tumor response to radiation or chemo-radiation combo.

DETAILED DESCRIPTION:
PHASE: II/III

OBJECTIVES:

Primary: To investigate the clinical value of serial quantitative [F-18] FLT positron image assessment of tumor proliferation rates for early assessment of tumor response to radiation or chemoradiotherapy regimens (except with 5-fluorouracil) in comparison to serial quantitative [F-18] FDG images

Secondary: To gain additional clinical information and experience with [F-18]FLT to guide the design of a future, pivotal, Phase III trial where changes in tumor proliferation from pre-treatment baseline values can be used as a early indicator of response to therapy regimens.

DESIGN: Open label, nonrandomized, uncontrolled, single group assignment

DURATION: Pre treatment [F-18] FLT PET scan following a clinical [F-18] FDG PET scan followed by post treatment [F-18] FLT PET scan and a post treatment, clinical [F-18] FDG PET scan at 4 weeks (±1 week) to monitor radiotherapy or chemoradiotherapy.

PROCEDURES: Informed consent, collection of demographic information, medical history, physical examinations, vital signs, 12-lead ECGs, concomitant medication collection, monitor adverse events, pre treatment [F-18] FLT PET scan and post treatment [F-18] FLT PET scan

SUBJECTS: Approximately 60 patients will be enrolled with confirmed lung cancer, or head and neck cancer. The patients must also be starting radiotherapy or a chemoradiotherapy regimen (except with 5-fluorouracil) to be eligible. This allows for approximately 40 evaluable patients to complete this study at approximately four to eight sites and conducted in the United States.

ELIGIBILITY:
Inclusion Criteria:

* Patient provides written Informed Consent and is willing to comply with protocol requirements
* Patient is at least 18 years of age on the day of dosing (male or female of any race or ethnicity)
* Patient is capable of lying still in the PET scanner for the protocol required time frame(s)
* Patient has a diagnosis of one of the following malignancies using the TNM Staging System:
* Lung cancer (T3 grade up, node positive, but no metastatic disease)
* Head and neck cancer (T3 grade up, node positive, but no metastatic disease)
* Patient has undergone a comparative, diagnostic procedure with lesion(s) visible, other than ultrasound, that includes, but is not limited to computed tomography (CT), magnetic resonance imaging (MRI), nuclear medicine imaging, endoscopy, laparoscopy, standard abdominal x-ray, biopsy and/or surgery for one of the above mentioned areas
* Patient is scheduled to start radiotherapy or a chemoradiotherapy regimen for curative intent
* As a part of his/her standard radiotherapy or chemoradiotherapy regimen, patient is scheduled to have clinical [F-18]FDG PET scans pre treatment and post treatment (at about 4 weeks (±1 week) after the start of therapy)
* Patient is scheduled to have the investigational, pre treatment [F-18] FLT PET scan recommended to be within ± 2 days of the clinical, pre treatment [F-18] FDG PET scan
* Patient has not received or intends to receive 5-fluorouracil (chemotherapeutic agent)
* Patient has a score of greater than or equal to (>/=) 60% on the Karnofsky Performance Status Scale

Exclusion Criteria:

* Patient is a pregnant or lactating female. Exclude the possibility of pregnancy:
* by testing on site at the institution (serum or urine βHCG) within 48 hours prior to the start of each investigational product administration
* by surgical history (eg, tubal ligation or hysterectomy)
* by patient's history of being post menopausal with a minimum 1 year without menses
* Patient is undergoing treatment with palliative intent
* Patient has received an investigational compound and/or medical device within 14 days before admission into this study
* Patient has any medical condition or other circumstances which would significantly decrease the chances of obtaining reliable data, achieving study objectives, or completing the study and/or post-dose follow-up examinations
* Patient is determined by the Investigator that he/she is clinically unsuitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2009-02; Primary Completion 2010-08 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ebrahim S Delpassand, MD, Principal Investigator — Excel Diagnostics Imaging Clinics; Michael Brandt-Zawadzki, MD, Principal Investigator — Hoag Memorial Hospital, Newport Beach, CA
Locations (2):
- United States (2):
  - Hoag Memorial Hospital, Newport Beach, California
  - Excel Diagnostics Imaging Clinics, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 49 patients were enrolled and 38 patients received investiational product.
Groups:
- [F-18]FLT PET Scan: Open label, nonrandomized, uncontrolled, single group assignment, multi-center clinical trial to evaluate [F-18] FLT as a PET imaging tool in cancer patients clinically scheduled for treatment with radiation or radiation - chemotherapy. Standard [F-18] FDG PET will be the active comparator.
Period: Overall Study
Arm/Group | [F-18]FLT PET Scan
Started | 49
Completed | 38
Not Completed | 11

BASELINE CHARACTERISTICS:
Population: A total of 49 patients were enrolled and 38 patients received investiational product.
Arm/Group | [F-18]FLT Scan
Number analyzed (Participants) | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 22
Age Continuous [Mean (Standard Deviation); unit: years] | 64.67 (10.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 23
Region of Enrollment [Number; unit: participants]
  United States | 49

OUTCOME MEASURES:

1. Primary Outcome: [F-18]FLT PET Scan for Early Assessment of Tumor Response to Radiation or Chemoradiotherapy Compared to [F-18] FDG PET Scan
Description: The sponsor decided not to further develop [F-18]FLT. Therefore, no further analysis was performed.
Time Frame: 3-5 weeks after the start of radiation or chemo radio therapy
Arm/Group | [F-18]FLT PET Scan
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 48 patients received investigational product at Visit 2 and 41 patients received investigational product at Visit 3
Description: 48 patients received any amount of investigational prduct. One patient experienced AE prior to receiving any investigational product and was therefore not included in the naalysis of AE and concomitant medications.
Arm/Group | [F-18]FLT PET Scan
Serious Adverse Events (participants affected / at risk) | 0/38
Other Adverse Events (participants affected / at risk) | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The restriction on the PI is that the sponsor can review results communication prior to public release and can embargo communications regarding trial results.